CLINICAL TRIAL: NCT04688853
Title: A Phase I Study to Investigate the Safety, Tolerability and Preliminary Efficacy of TEG002 Infusion in Relapsed/Refractory Multiple Myeloma Patients
Brief Title: A Study to Investigate the Safety and Efficacy of TEG002 in Relapsed/Refractory Multiple Myeloma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gadeta B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TEG002_MM_US_01
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma, Refractory; Multiple Myeloma in Relapse; Multiple Myeloma
Keywords: T cell therapy; Engineered T Cells; TEG; TEGs; TEG002
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm, Open label (Experimental): This is a single arm, open-label, multicenter phase I study with a dose escalation and an expansion segment.
  For the Dose escalation segment, 3-9 patients per dose cohort will receive:
  * Dose level 1: Low
  * Dose level 2: Medium
  * Dose level 3: High
  For the expansion segment, additional patients may be enrolled until a maximum of 20 patients have received the recommended dose
  Interventions: Biological: TEG002

INTERVENTIONS:
Biological: TEG002 — TEG002 cells are autologous T cells transduced with a specific γδTCR

SUMMARY:
This is a single arm, open-label, multicenter phase I study to assess the safety, tolerability and preliminary efficacy of autologous T cells transduced with a specific γδTCR, i.e. TEG002, in a dose escalation and expansion study in relapsed/refractory Multiple Myeloma patients.

The study will comprise of a Dose Escalation Segment and an Expansion Segment. The study consists of a screening period, leukapheresis of mononuclear cells, and conditioning chemotherapy, followed by TEG002. All subjects continue to be followed regularly for safety and efficacy assessments until 1 year after TEG002 administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adult
* Relapsed or refractory Multiple Myeloma as defined by the IMWG
* Life expectancy ≥3 months
* ECOG performance status 0 or 1
* Adequate vital organ function
* Adequate bone marrow function
* Toxicities from prior/ongoing therapies recovered to ≤ Grade 2 or subject's baseline
* WCBP and men who can father children must be willing and able to use adequate contraception

Exclusion Criteria:

* Any uncontrolled medical or psychiatric disorder that would preclude participation as outlined
* Pregnant or lactating women
* Amyloidosis
* Uncontrolled infection(s)
* Active CNS disease
* Previous allogeneic-HSCT
* History of another primary malignancy that requires intervention beyond surveillance or that has not been in remission for at least 1 year.
* Subjects that received experimental or systemic therapy < 14 days before TEG002 infusion
* NYHA Class ≥ II
* Patients depending on dialysis
* Patients with a history of pulmonary embolism or deep vein thrombosis
* T cell mediated active autoimmune disease OR any active autoimmune disease requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Safety determined by incidence of (S)AEs by type and grade, including the occurrence of dose-limiting toxicities (DLTs) | Until day 28 following infusion
  For the dose escalation segment: Safety determined by incidence of (S)AEs by type and grade, including the occurrence of dose-limiting toxicities (DLTs)
Safety: For the expansion segment: Confirmation of safety determined by the incidence of (S)AEs by type and grade | Until year 2
  For the expansion segment: Confirmation of safety determined by the incidence of (S)AEs by type and grade

SECONDARY OUTCOMES:
Feasibility of TEG002 generation in r/r MM patients as measured by the number of TEG002 products successfully generated in r/r MM patients | Assessment per subject production run, timeframe: prior to day 0 for each subject
  Feasibility of TEG002 generation in r/r MM patients as measured by the number of TEG002 products successfully generated in r/r MM patients
TEG002 efficacy by looking at Objective response rate | Until Year 2
  Efficacy: Objective response rate
TEG002 efficacy by looking at Overall survival | Until Year 2
  Efficacy: Overall survival
TEG002 efficacy by looking at Progression free survival | Until Year 2
  Efficacy: Progression free survival
TEG002 efficacy by looking at Duration of response | Until Year 2
  Efficacy: Duration of response
TEG002 efficacy by looking at Time to response | Until Year 2
  Efficacy: Time to response
TEG002 efficacy by looking at Time to progression | Until Year 2
  Efficacy: Time to progression
TEG002 pharmacokinetics measured in blood in bone marrow over time | Until Year 2
  Safety & Efficacy: TEG002 persistence measured by qPCR in blood in bone marrow over time
TEG002 pharmacodynamics as measured by IL6 level in serum over time | until Year 2
  Safety & Efficacy: TEG002 pharmacodynamics measured by the level of IL6 in serum over time
TEG002 pharmacodynamics as measured by CRP level in serum over time | until Year 2
  Safety & Efficacy: TEG002 pharmacodynamics measured by the CRP level in serum over time
TEG002 pharmacodynamics as measured by ferritin level in serum over time | until Year 2
  Safety & Efficacy: TEG002 pharmacodynamics measured by the ferritin level in serum over time

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts